CLINICAL TRIAL: NCT06431048
Title: No DIET Trial: Dogmatic Interruption of Enteral nuTrition
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Jeffrey Coughenour (Other)
Responsible Party: Sponsor-Investigator, Jeffrey Coughenour, Associate Professor of Clinical Surgery, University of Missouri-Columbia
Organization: University of Missouri-Columbia (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2101744
Record Dates: First submitted 2024-05-16; First posted 2024-05-28 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Gastrostomy; Tracheostomy
Keywords: Percutaneous Endoscopic Gastrostomy; Tracheostomy; Enteral feeding

STUDY DESIGN:
Intervention Model Description: The two groups per arm in this study are:
  1. Nutrition will be stopped when the patient is called to the OR for scheduled procedure.
  2. Nutrition will be stopped 2 hours before the scheduled procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients receiving PEG nutrition, scheduled for tracheostomy placement. (Experimental)
  Interventions: Other: Naso-enteral nutrition will be stopped when the patient is called to the OR for scheduled procedure.; Other: Naso-enteral nutrition will be stopped 2 hours before the scheduled procedure.
- Patients receiving naso-enteral feeding, scheduled for PEG placement. (Experimental)
  Interventions: Other: Naso-enteral nutrition will be stopped when the patient is called to the OR for scheduled procedure.; Other: Naso-enteral nutrition will be stopped 2 hours before the scheduled procedure.

INTERVENTIONS:
Other: Naso-enteral nutrition will be stopped when the patient is called to the OR for scheduled procedure. — Naso-enteral nutrition will be stopped when the patient is called to the OR for scheduled procedure (tracheostomy + PEG or PEG only).
Other: Naso-enteral nutrition will be stopped 2 hours before the scheduled procedure. — Naso-enteral nutrition will be stopped 2 hours before the scheduled procedure (tracheostomy + PEG or PEG only).

SUMMARY:
There is currently limited guidance on when to hold nutritional supplementation through for patients, who are receiving tube feeding, undergoing surgical procedures. This study aims to investigate which time would be the best to stop nutrition, if at all, before undergoing a surgical procedure.

DETAILED DESCRIPTION:
The risk for malnutrition-associated complications is high for patients in the trauma- surgical-, and neurological intensive care units. Patients with persistent neurologic impairment often require nutritional supplementation through a variety of naso-enteral or surgical feeding tubes such as percutaneous endoscopic gastrostomy (PEG) tubes. In patients with a protected airway, enteral nutrition has been reported to continue during invasive surgical procedures. Nonetheless, University Hospital's current SOC for holding enteral nutrition prior to undergoing surgical procedures under anesthesia is 8 hours. However, the current American Society of Anesthesiologists (ASA) guidelines do not make provision for inpatients receiving supplemental enteral nutrition. Enteral nutrition contains protein, fat, and carbohydrates, mimicking what patients would consume with a solid food meal. Balancing the need of optimized nutrition in critically ill patients with an unprotected airway against the risk of aspiration during surgical procedures brings a need for clear guidance on when to hold enteral nutrition prior to undergoing a tracheostomy procedure.

ELIGIBILITY:
Inclusion criteria:

* Patients aged >18 years.
* Patients who require a tracheostomy or PEG placement.

Exclusion criteria:

* Patients with gastric and/or bowel obstruction.
* Patients unable to receive enteral nutrition.
* Patients who are pregnant and/or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-06-25 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Measuring stomach contents in patients undergoing a tracheostomy and/or PEG placement. | 0-8 hours
  Measurement of stomach contents will be done with enteral feeding stopped at different time points prior to undergoing the surgical procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Coughenour, MD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri Hospital, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Glanz, S. Hold the feeds … or not? Exploring intraoperative feeding. Published online 2019:2017-2019.
- [Background] Practice Guidelines for Preoperative Fasting and the Use of Pharmacologic Agents to Reduce the Risk of Pulmonary Aspiration: Application to Healthy Patients Undergoing Elective Procedures: An Updated Report by the American Society of Anesthesiologists Task Force on Preoperative Fasting and the Use of Pharmacologic Agents to Reduce the Risk of Pulmonary Aspiration. Anesthesiology. 2017 Mar;126(3):376-393. doi: 10.1097/ALN.0000000000001452. No abstract available. PMID 28045707
- [Background] Carmichael H, Joyce S, Smith T, Patton L, Lambert Wagner A, Wiktor AJ. Safety and efficacy of intraoperative gastric feeding during burn surgery. Burns. 2019 Aug;45(5):1089-1093. doi: 10.1016/j.burns.2018.12.009. Epub 2019 Apr 1. PMID 30948280
- [Background] Schneider JA, Lee YJ, Grubb WR, Denny J, Hunter C. Institutional practices of withholding enteral feeding from intubated patients. Crit Care Med. 2009 Jul;37(7):2299-302. doi: 10.1097/CCM.0b013e3181a007eb. PMID 19455023
- [Background] Shahmanyan D, Lawrence JC, Lollar DI, Hamill ME, Faulks ER, Collier BR, Chestovich PJ, Bower KL. Early feeding after percutaneous endoscopic gastrostomy tube placement in patients who require trauma and surgical intensive care: A retrospective cohort study. JPEN J Parenter Enteral Nutr. 2022 Jul;46(5):1160-1166. doi: 10.1002/jpen.2303. Epub 2022 Jan 27. PMID 34791680